CLINICAL TRIAL: NCT00711451
Title: Manual and Expressed Placental Removal at Planned Cesarean Delivery and Its Effects on Various Cardiac Indices as Measured By Continuous Wave Doppler Ultrasonography
Brief Title: Manual and Expressed Placental Removal at Cesarean Delivery and Its Effects on Various Cardiac Indices
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: unable to recruit patients
Sponsor: Corewell Health East (Other)
Responsible Party: Principal Investigator, John Uckele, Attending Physician, Corewell Health East
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2008-056
Record Dates: First submitted 2008-07-02; First posted 2008-07-08 (Estimated); Last update posted 2012-07-16 (Estimated); Status verified 2012-07

CONDITIONS: Pregnancy; Cesarean Delivery
Keywords: systemic vascular resistance; pregnancy; scheduled cesarean delivery; syncytiotrophoblast apoptosis; continuous wave Doppler
MeSH Terms: interventions — Gene Expression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- manual (Active Comparator): Manual removal of placenta
  Interventions: Behavioral: Manual removal
- expressed (Active Comparator): expressed placental removal
  Interventions: Procedure: Expressed removal

INTERVENTIONS:
Behavioral: Manual removal — Manual removal of placenta during cesarean delivery
  Other Names: manual
  Arms: manual
Procedure: Expressed removal — Surgeon will perform an expressed delivery of the placenta
  Other Names: expressed
  Arms: expressed

SUMMARY:
The purpose of this study is to evaluate whether manual removal of the placenta during a cesarean delivery results in higher changes in the resistance of blood flow throughout the body, also called systemic vascular resistance (SVR)

DETAILED DESCRIPTION:
Patients presenting to William Beaumont Hospital Royal Oak Labor and Delivery for a scheduled low transverse cesarean delivery will be asked to participate in a prospective, randomized study to evaluate any changes in systemic vascular resistance (SVR) pre- and post-delivery.

After obtaining informed consent, the patients will be randomized to one of two groups: group 1 will have manual removal of the placenta at cesarean section and group 2 will have expressed removal of the placenta at cesarean section.

Both groups will have a pre-operative continuous wave Doppler evaluation and a post-operative continuous wave Doppler evaluation at 24 hours after delivery. Continuous wave Doppler evaluation will be used pre- and post-operatively to evaluate any changes in SVR.

ELIGIBILITY:
Inclusion Criteria:

* pregnant
* scheduled for cesarean delivery
* able to give informed consent

Exclusion Criteria:

* taking medications that may affect hemodynamics
* unable to give informed consent

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2008-07; Primary Completion 2011-02 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Hemodynamic profile, especially Systemic Vascular Resistance | immediately before and 24 hours after cesarean delivery

SECONDARY OUTCOMES:
development of postpartum preeclampsia | within 1 week of delivery

CONTACTS AND LOCATIONS:
Overall Officials: Christian Bogner, MD, Principal Investigator — Corewell Health East
Locations (1):
- William Beaumont Hospital, Royal Oak, Michigan, United States